CLINICAL TRIAL: NCT07290322
Title: Denture Retention of Intra-orally Scanned Versus Extra-orally Scanned Digitally Printed Maxillary Denture in Completely Edentulous Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rehab Rabie Abdalla, Masters student, Cairo University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21-12-2023
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Complete Edentulism
Keywords: Intraoral scanning; Extra oral scaning; Complete edentulism; Digital; denture retention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-Orally Scanned Dentures (Experimental): Participants in this arm will recieve maxillary dentures fabricated using intraoral scanning technology . digital impressions of the oral cavity will be captured directly using the 3 shape trios intraoral scanner, eliminating the need for conventional impression materials , these digital impressions will be used to design and 3D print the dentures , which will then be fitted and evaluated for retention .
  Interventions: Device: extraorally scanned methods
- Extra-Orally Scanned Dentures (Active Comparator): Participants in this arm will recieve maxillary dentures fabricated using extraoral scanning technology . conventional impressions of the oral cavity will first be taken using traditional impression material , these impressions will then be scanned externally using the 3Shape scanner to create digital models . these digital models will be used to design and 3D print the dentures , which will then be fitted and evaluated for retention .
  Interventions: Device: Intaorally scanned methods

INTERVENTIONS:
Device: Intaorally scanned methods — the intraoral scanning method involves capturing digital impressions of the oral cavity directly using the 3 shape scanner . this method eliminates the need for traditional impression material providing a more comfortable and precise imaging process , the digital impressions are the utilized to design and fabricate maxillary dentures using 3D printing technology . the intervention focuses on evaluating denture's retention
  Arms: Extra-Orally Scanned Dentures
Device: extraorally scanned methods — The extra-oral scanning method involves creating conventional impressions of the oral cavity using traditional impression materials. These impressions are then scanned externally using the 3Shape scanner to produce digital models. The digital models are used to design and fabricate maxillary dentures through 3D printing technology. This intervention aims to assess denture retention
  Arms: Intra-Orally Scanned Dentures

SUMMARY:
The goal of this clinical trial is to evaluate denture retention in intra-orally scanned versus extra-orally scanned digitally printed maxillary dentures in completely edentulous patients. The main question is : 1. Do intra-orally scanned dentures provide better retention compared to extra-orally scanned dentures? Researchers will compare the intra-orally scanned denture group to the extraorally scanned denture group to determine if one method leads to superior retention records.

Participants will:

• Receive both types of dentures (intra-orally scanned and extra-orally scanned), with a three-week wash-out period between each intervention. The study aims to provide evidence on the optimal scanning method for digitally printed maxillary dentures in edentulous patients.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate and compare denture retention with intra-orally scanned and extra-orally scanned digitally printed maxillary dentures in completely edentulous patients. This in vivo study seeks to provide insights into how the scanning method impacts the comfort, fit, and retention of maxillary dentures, ultimately guiding clinicians in choosing the most patient preferred approach.

Study Design and Objectives This study involves eight completely edentulous participants who will receive both types of dentures-one set based on intra-oral scanning and another based on extra-oral scanning. A wash-out period of two weeks between the use of each denture ensures that the effects of one intervention do not influence the results of the other. The primary objective of this study are:

1. To determine if intra-orally scanned dentures provide higher denture retention compared to extra-orally scanned dentures.

Study Methodology

Participants will undergo the following steps:

1. Scans and Fabrication:

   * Intra-oral scanning will be performed using the 3Shape scanner to capture precise digital impressions of the oral cavity.
   * For the extra-oral scanning, conventional impressions will first be taken, and these will be scanned externally using the same scanner to create digital models.
   * Both types of digital models will be used to fabricate maxillary dentures using 3D printing technology.
2. Fitting and Wash-out Period:

   * Participants will first use one type of denture (either intra-oral or extra-oral scanned) for a designated period.
   * After a two-week wash-out period without wearing dentures, they will switch to the other type of denture.
3. Data Collection:

   * After wearing each type of denture, participants will complete be exposed to The assessment of denture retention which involves measuring the force required to dislodge the denture in different directions .

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous patients
* Angle's class I Skeletal relationship
* normal facial symmetry
* comparative patients

Exclusion Criteria:

* tempromandibular disorders
* uncontrolled diabetes
* patients with neuromuscular disorders
* severe psychiatric disorders
* angle's class II and III skeletal relationship

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Denture Retention | the patient is observed for three weeks as awash_out period after each type of scan so that i can compare the denture retention across those periods

CONTACTS AND LOCATIONS:
Overall Officials: Rehab R Abdalla, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
At this time, no final decision has been made regarding the sharing of IPD. We will consider sharing the data based on ethical guidelines and the research objectives in the future.

REFERENCES:
- [Result] 1-Comparative Accuracy of Intraoral and Extraoral Digital Scanners by MA Mansoor et al., published in the Journal of Prosthetic Dentistry in 2024. 2.The Accuracy of Intraoral Scan in Obtaining Digital Impressions of Edentulous Jaws by Y Wang et al., published in the Journal of Prosthetic Dentistry in 2024. 3.Comparison of Intraoral and Extraoral Digital Scanners: Evaluation of Surface Topography and Precision, published on ResearchGate in 2020. 4.Effect of Different Scanning Protocols on the Retention of Complete Dentures by SM Fadl et al., published in the Egyptian Dental Journal in 2023.
- See also: This study, titled "Effect of Different Scanning Protocols on the Retention of Duplicated Maxillary Complete Dentures," investigates how various scanning techniques influence the retention and fit of maxillary complete dentures. It provides insights into — https://edj.journals.ekb.eg/article_320095_3b8d81bc7d4bfd02956352980006502d.pdf?utm_source=chatgpt.com